CLINICAL TRIAL: NCT03416855
Title: A Multi-centre, Prospective, Open-label, Single-arm, Non-interventional, Regulatory Post Marketing Surveillance(rPMS) Study of Ryzodeg® FlexTouch® (Insulin Degludec /Insulin Aspart) to Evaluate Safety and Effectiveness in Patients With Diabetes Mellitus in Routine Clinical Practice in Korea
Brief Title: A Regulatory Post Marketing Surveillance (rPMS) Study of Ryzodeg® FlexTouch® (Insulin Degludec /Insulin Aspart) to Evaluate Safety and Effectiveness in Patients With Diabetes Mellitus in Routine Clinical Practice in Korea
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN5401-4196; 1111-1194-8505 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overall population: Participants will be decided to be treated with Ryzodeg® FlexTouch® by physicians before the enrolment in the study based on clinical judgement in the diabetes management.
  Interventions: Drug: Insulin degludec /insulin aspart

INTERVENTIONS:
Drug: Insulin degludec /insulin aspart — Commercially available Insulin degludec /insulin aspart (Ryzodeg® FlexTouch®) according to routine clinical practice at the discretion of the treating physician.
  Other Names: Ryzodeg® FlexTouch®

SUMMARY:
The purpose of this study is to collect information about safety and effectiveness of Ryzodeg® FlexTouch® in participants with diabetes mellitus requiring insulin therapy under routine clinical practice conditions with the aim of identifying or quantifying a safety hazard, early detection of unknown safety problems. Participants will attend the clinic/hospital/medical institution according to usual practice and receive medical care, as agreed with the study doctor.

ELIGIBILITY:
Inclusion Criteria: - The decision to initiate treatment with commercially available Ryzodeg® FlexTouch® has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study - Signed informed consent obtained before any study related activities. Study related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study - Age equals to or more than 2 years at the time of signing informed consent with diabetes mellitus (Type 1 or Type 2) and who is scheduled to start treatment with Ryzodeg® FlexTouch® based on the clinical judgment of their treating physician as specified in the Korean-Prescribing information (K-PI) Exclusion Criteria: - Patients who are or have previously been on Ryzodeg® FlexTouch® therapy - Known or suspected hypersensitivity to Ryzodeg® FlexTouch®, the active substance or any of the excipients - Previous participation in this study. Participation is defined as having given informed consent in this study - Female patient who is pregnant, breast-feeding or intends to become pregnant and is of childbearing potential and not using adequate contraceptive methods(adequate contraceptive measures as required by Korea regulation or practice) - Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diabetes mellitus, who are scheduled to start treatment with Ryzodeg® FlexTouch® based on the clinical judgment of their treating physician as specified in the Korean-Prescribing information
Sampling Method: Non-Probability Sample
Enrollment: 768 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-05-19 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events (AEs) at week 13 | week 13 (± 2 weeks)
  Count of events
Number of patients with AEs at week 13 | week 13 (± 2 weeks)
  Number of patients
Percentage of patients with AEs at week 13 | week 13 (± 2 weeks)
  Percentage of patients
Number of Adverse events (AEs) at week 26 | week 26 (± 2 weeks)
  Count of events
Number of patients with AEs at week 26 | week 26 (± 2 weeks)
  Number of patients
Percentage of patients with AEs at week 26 | week 26 (± 2 weeks)
  Percentage of patients

SECONDARY OUTCOMES:
Number of patients with Adverse Drug Reaction (ADR) at week 13 | week 13 (± 2 weeks)
  Number of patients
Percentage of Patients with ADR at week 13 | week 13 (± 2 weeks)
  Percentage of patients
Number of Patients with ADR at week 26 | week 26 (± 2 weeks)
  Number of patients
Percentage of Patients with ADR at week 26 | week 26 (± 2 weeks)
  Percentage of patients
Number of patients with Serious AE/ADR at week 13 | week 13 (± 2 weeks)
  Number of patients
Percentage of patients with Serious AE/ADR at week 13 | week 13 (± 2 weeks)
  Percentage of patients
Number of patients with Serious AE/ADR at week 26 | week 26 (± 2 weeks)
  Number of patients
Percentage of patients with Serious AE/ADR at week 26 | week 26 (± 2 weeks)
  Percentage of patients
Number of patients with unexpected ADR at week 13 | week 13 (± 2 weeks)
  Number of patients
Percentage of patients with unexpected ADR at week 13 | week 13 (± 2 weeks)
  Percentage of patients
Number of subjects with unexpected ADR at week 26 | week 26 (± 2 weeks)
  Number of subjects
Percentage of patients with unexpected ADR at week 26 | week 26 (± 2 weeks)
  Percentage of patients
Number of patients with Severe or Blood Glucose (BG) confirmed hypoglycaemia (Plasma Glucose <56 mg/dl) at week 13 | week 13 (± 2 weeks)
  Number of patients
Percentage of patients with Severe or BG confirmed hypoglycaemia (Plasma Glucose <56 mg/dl) at week 13 | week 13 (± 2 weeks)
  Percentage of patients
Number of patients with Severe or BG confirmed hypoglycaemia (Plasma Glucose <56 mg/dl) at week 26 | week 26 (± 2 weeks)
  Number of patients
Percentage of patients with Severe or BG confirmed hypoglycaemia (Plasma Glucose <56 mg/dl) at week 26 | week 26 (± 2 weeks)
  Percentage of patients
Change from baseline in body weight at week 13 | week 0, week 13 (± 2 weeks)
  Measured in kg
Change from baseline in body weight at week 26 | week 0, week 26 (± 2 weeks)
  Measured in kg
Insulin dose at week 13 | week 13 (± 2 weeks)
  Dose in Units
Insulin dose at week 26 | week 26 (± 2 weeks)
  Dose in Units
Change from baseline in HbA1c after 13 weeks of treatment | week 0, week 13 (± 2 weeks)
  Measured in %
Change from baseline in HbA1c after 26 weeks of treatment | week 0, week 26 (± 2 weeks)
  Measured in %
Percentage of patients achieving the target of HbA1c < 7.0% at 13 weeks of treatment | week 13 (± 2 weeks)
  Percentage of patients
Percentage of patients achieving the target of HbA1c < 7.0% at 26 weeks of treatment | week 26 (± 2 weeks)
  Percentage of patients
Change from baseline in Fasting Blood Glucose/Plasma Glucose (FBG/FPG) after 13 weeks treatment | week 0, week 13 (± 2 weeks)
  Measured in mg/dl or other equivalent SI units
Change from baseline in FBG/FPG after 26 weeks treatment | week 0, week 26 (± 2 weeks)
  Measured in mg/dl or other equivalent SI units
Changes from baseline in Post Prandial Blood/Plasma Glucose (PPBG/PPPG) after 13 weeks treatment | week 0, week 13 (± 2 weeks)
  Measured in mg/dl or other equivalent SI units
Changes from baseline in PPBG/PPPG after 26 weeks treatment | week 0, week 26 (± 2 weeks)
  Measured in mg/dl or other equivalent SI units

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (13):
- South Korea (13):
  - Novo Nordisk Investigational Site, Busan
  - Novo Nordisk Investigational Site, Daegu
  - Novo Nordisk Investigational Site, Daejeon
  - Novo Nordisk Investigational Site, Gangwon-do
  - Novo Nordisk Investigational Site, Goyang
  - Novo Nordisk Investigational Site, Gyeonggi-do
  - Novo Nordisk Investigational Site, Incheon
  - Novo Nordisk Investigational Site, Jeonju
  - Novo Nordisk Investigational Site, Pusan
  - Novo Nordisk Investigational Site, Seoul
  - Novo Nordisk Investigational Site, Suwon
  - Novo Nordisk Investigational Site, Suwon-si, Gyeonggi-do
  - Novo Nordisk Investigational Site, Ulsan

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://www.novonordisk-trials.com/website/content/how-to-access-clinical-trial-datasets.aspx